CLINICAL TRIAL: NCT05355090
Title: Effects of Daily Protein Supplementation for 8 Weeks on Improved Glucose, Insulin, and HbA1c Levels in Pre-Diabetics or Type 2 Diabetes Mellitus
Brief Title: Daily Protein Pacing Effects on HbA1c in Type 2 Diabetics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2111-1004
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes; HbA1c; Protein Intake
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 24 volunteers with pre-diabetes or Type 2 diabetes mellitus (n=24) will be quasi-randomized to one of the two groups matched by sex (men/women) and body weight. Participants will be enrolled in the study as a single cohort and participate in a 8-week protein supplementation regimen consisting of three daily servings of whey protein along with their typical dietary intake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein Pacing (Experimental): During the 8 week trial, the Protein Pacing (PP) group will consume 3 daily servings of whey protein powder mixed with water at timed intervals: morning (0600-0800), afternoon (1000-1400), and evening (2000-2200) in addition to their normal food intake.
  Interventions: Dietary Supplement: PP
- Standard Diet (No Intervention): The participants in the CON will continue with their usual habitual dietary intake over the 8-week study and receive no intervention.

INTERVENTIONS:
Dietary Supplement: PP — Protein Pacing three times per day
  Arms: Protein Pacing

SUMMARY:
This study will examine the effects of protein (whey) supplementation added to the normal diet of pre-diabetes or diagnosed type 2 diabetes mellitus (T2DM) men and women on plasma glycated hemoglobin (HbA1c) and total body fat levels. Specifically, this study will directly quantify the impact of 3x/day timed ingestion of supplemental whey protein (20 grams of 80 calories per serving) added to the normal diet of free-living pre-diabetic or T2DM men and women over an 8-week study period on the major diagnostic outcome of pre-diabetic and T2DM (HbA1c levels) and total body fat levels. This study will quantify changes in HbA1C and total body fat levels in 24 pre-diabetics or T2DM participants.

DETAILED DESCRIPTION:
Previous investigations have demonstrated that simply adding 3 small protein feedings to the normal diet of overweight men and women, independent of caloric restriction and/or engaging in exercise training, significantly reduces body weight, fat mass, abdominal fat, waist circumference, and blood fat (triglyceride) levels (Arciero et al JAP, 2014), and confirms previous research (Baer et al, J Nutr, 2011). This timed ingestion is referred to as protein pacing (PP) and has been utilized in numerous scientific investigations with a great deal of success by the PI (see references). This one, simple, dietary modification, independent of reducing calorie intake and/or engaging in exercise training, is noteworthy and exceptional in terms of health improvements derived from diet alone. Unfortunately, the incidence and healthcare costs associated with type 2 diabetes mellitus (T2DM) are overwhelming. Currently, more than 34 million Americans have T2DM (1 in 10) and is increasing at alarming rates (>4.0%/year) among all segments of the population. Equally disturbing, T2DM costs the US more than $330 billion a year, including $237 billion in direct medical costs and $90 billion in reduced worker productivity. Thus, identifying evidence-based, effective, time-efficient, and easy-to-follow lifestyle strategies are vital to reducing these staggering healthcare costs and improving the health of T2DM patients. Indeed, lifestyle therapies remain the most effective treatments for T2DM outcomes.

The purpose of this study is to examine the effects of protein (whey) supplementation added to the normal diet of pre-diabetes or diagnosed type 2 diabetes mellitus (T2DM) men and women on plasma glycated hemoglobin (HbA1c) and total body fat levels. Specifically, this study will directly quantify the impact of 3x/day timed ingestion of supplemental whey protein (20 grams of 80 calories per serving) added to the normal diet of free-living pre-diabetic or T2DM men and women over an 8-week study period on the major diagnostic outcome of pre-diabetic and T2DM (HbA1c levels) and total body fat levels. This study will quantify changes in HbA1C and total body fat levels in 24 pre-diabetics or T2DM participants.

ELIGIBILITY:
Inclusion Criteria:

* non-smoker
* weight stable (+/-2kg) for at least 6 months prior to beginning the study
* Pre-diabetic and Type 2 diabetic mellitus men and women with no known significant cardiovascular or metabolic diseases as assessed by a medical history and a comprehensive medical examination by their physicians
* Sedentary or lightly active (<30 min, 2d/wk of structured physical activity) as assessed by a Physical Activity questionnaire

Exclusion Criteria:

* Emphysema
* Significant heart disease (CABG, CHF, VFib, Hypercholesterolemia, Uncontrolled High Blood Pressure, etc.)
* COPD
* Cancer or undergoing treatment for cancer
* Allergies to milk or milk products, sugar alcohols, fructose, or gluten
* Anorexia or Bulimia
* Fasting intolerances/hypoglycemia
* pregnant women or those looking to become pregnant

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 0 and 4, and 8 weeks
  Quantify changes in HbA1c blood levels vja finger stick of 40ul or venipuncture blood draw of 5ml per visit (weeks 0, 4, and 8)

SECONDARY OUTCOMES:
Change in total body fat and lean body mass | 0, 4 and 8 weeks
  Quantitative measure of total body fat and muscle mass in kilograms using BODPod (air displacement plethysmography
Change in blood glucose, and lipids | 0, 4 and 8 weeks
  Finger stick of 40ul or venipuncture blood draw of 5ml per visit (weeks 0, 4, and 8) to quantify changes in mg/dL
Change in physical activity | 0, 4, and 8 weeks
  Quantitative measure of physical activity (kilocalories per day) using the ActiGraph accelerometer
Change in body weight | weeks 0, 4, and 8
  Quantitative measure of body weight in kilograms using a standard scale

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Arciero, PhD, Principal Investigator — Skidmore College
Locations (1):
- Human Nutrition and Metabolism Laboratory, Saratoga Springs, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arciero PJ, Edmonds R, He F, Ward E, Gumpricht E, Mohr A, Ormsbee MJ, Astrup A. Protein-Pacing Caloric-Restriction Enhances Body Composition Similarly in Obese Men and Women during Weight Loss and Sustains Efficacy during Long-Term Weight Maintenance. Nutrients. 2016 Jul 30;8(8):476. doi: 10.3390/nu8080476. PMID 27483317
- [Background] Arciero PJ, Baur D, Connelly S, Ormsbee MJ. Timed-daily ingestion of whey protein and exercise training reduces visceral adipose tissue mass and improves insulin resistance: the PRISE study. J Appl Physiol (1985). 2014 Jul 1;117(1):1-10. doi: 10.1152/japplphysiol.00152.2014. Epub 2014 May 15. PMID 24833780
- [Background] Arciero PJ, Ormsbee MJ, Gentile CL, Nindl BC, Brestoff JR, Ruby M. Increased protein intake and meal frequency reduces abdominal fat during energy balance and energy deficit. Obesity (Silver Spring). 2013 Jul;21(7):1357-66. doi: 10.1002/oby.20296. Epub 2013 May 23. PMID 23703835